CLINICAL TRIAL: NCT01370603
Title: A Randomized, Double-Blind, Active-Controlled, Multicenter, Crossover Study to Evaluate the Efficacy of Ezetimibe/Atorvastatin 10 mg/40 mg Fixed-Dose Combination Tablet Compared to Co-Administration of Marketed Ezetimibe 10 mg and Atorvastatin 40 mg in Patients With Primary Hypercholesterolemia
Brief Title: A Study to Evaluate the Effectiveness of Ezetimibe/Atorvastatin 10 mg/40 mg Combination Tablet Compared to Marketed Ezetimibe 10 mg and Atorvastatin 40 mg Tablets in Participants With High Cholesterol (MK-0653C-190 AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0653C-190
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; Ezetimibe; liptruzet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe and atorvastatin (Active Comparator): Medication will be administered in a double dummy fashion as 3 tablets orally on a daily basis, including 10 mg ezetimibe, 40 mg atorvastatin, and placebo to ezetimibe/atorvastatin.
  Interventions: Drug: Atorvastatin; Drug: Ezetimibe; Drug: Placebo to ezetimibe/atorvastatin
- Ezetimibe/atorvastatin combination (Experimental): Medication will be administered in a double dummy fashion as 3 tablets orally on a daily basis, including ezetimibe/atorvastatin 10 mg/40 mg, placebo to ezetimibe, and placebo to atorvastatin.
  Interventions: Drug: Ezetimibe/atorvastatin; Drug: Placebo to atorvastatin; Drug: Placebo to ezetimibe

INTERVENTIONS:
Drug: Atorvastatin — 40 mg tablet administered orally once daily
  Other Names: Lipitor®
  Arms: Ezetimibe and atorvastatin
Drug: Ezetimibe — 10 mg tablet administered orally once daily
  Other Names: Zetia®
  Arms: Ezetimibe and atorvastatin
Drug: Ezetimibe/atorvastatin — Ezetimibe/atorvastatin 10 mg/40 mg combination tablet administered orally once daily
  Other Names: Liptruzet®; MK-0653C
  Arms: Ezetimibe/atorvastatin combination
Drug: Placebo to atorvastatin — Administered orally once daily
  Arms: Ezetimibe/atorvastatin combination
Drug: Placebo to ezetimibe — Administered orally once daily
  Arms: Ezetimibe/atorvastatin combination
Drug: Placebo to ezetimibe/atorvastatin — Administered orally once daily
  Arms: Ezetimibe and atorvastatin

SUMMARY:
The purpose of this study is to determine whether ezetimibe/atorvastatin 10 mg/40 mg combination tablet is equivalent to the coadministration of ezetimibe 10 mg and atorvastatin 40 mg in lowering low-density-lipoprotein-cholesterol (LDL-C) after 6 weeks of treatment.

ELIGIBILITY:
Inclusion criteria:

* At low, moderate, or moderately high cardiovascular risk (according to National Cholesterol Education Program adult treatment panel III [NCEP ATP III] guidelines) and either statin-naïve with LDL-C ≥130 mg/dL for low risk or ≥100 mg/dL for moderate or moderately high risk OR on an allowable statin with on-therapy LDL-C ≥100 mg/dL in acceptable range and can safely discontinue and switch to study medication.
* Is willing to maintain a cholesterol-lowering diet throughout the study.
* Female of reproductive potential agrees to remain abstinent or to use (or have their partner use) 2 acceptable methods of birth control throughout the study.
* Female receiving non-cyclical hormone therapy, if maintained on a stable dose and regimen for at least 8 weeks prior to the study and if willing to continue the same regimen throughout the study.
* Off-therapy LDL-C levels are: for low risk patients, ≥130 mg/dL and ≤300 mg/dL; for moderate risk patients, ≥100 mg/dL and ≤300 mg/dL; for moderately high risk patients, ≥100 mg/dL and ≤275 mg/dL.
* Has liver transaminases ≤2 X upper limit of normal (ULN) with no active liver disease.
* Has creatine kinase (CK) levels ≤3 X ULN.
* Has triglyceride (TG) concentrations ≤400 mg/dL.

Exclusion criteria:

* Hypersensitivity or intolerance to ezetimibe, atorvastatin, the ezetimibe/atorvastatin combination tablet, or any component of these medications, or a history of myopathy or rhabdomyolysis with ezetimibe or any statin.
* Routinely consumes more than 2 alcoholic drinks per day (average >14 alcoholic drinks per week).
* Is pregnant or lactating.
* Has been treated with any other investigational drug within 30 days of the study.
* Is high risk (according to NCEP ATP III guidelines), including but not limited to one or more of the following: diabetes mellitus (Type I or II), myocardial infarction, coronary artery bypass surgery, angioplasty, stable or unstable angina.
* Has any of the following medical conditions: congestive heart failure; uncontrolled cardiac arrhythmias or recent significant changes in an electrocardiogram (ECG); homozygous familial hypercholesterolemia or has undergone LDL apheresis; partial ileal bypass, gastric bypass, or other significant intestinal malabsorption; uncontrolled hypertension; kidney disease; disease known to influence serum lipids or lipoproteins; hematologic, digestive, or central nervous system disorder; known to be human immunodeficiency virus (HIV) positive; history of malignancy ≤5 years prior to the study, except for adequately treated basal cell or squamous cell skin cancer or in situ

cervical cancer; mental instability, drug/alcohol abuse within the past 5 years, or major psychiatric illness not adequately controlled and stable on pharmacotherapy.

- Taking prohibited medications/foods including: systemic azole antifungals (e.g., fluconazole, ketoconazole), erythromycin or clarithromycin, and cyclosporine; ritonavir and saquinavir or lopinavir; >5 cups of grapefruit juice per day; combination therapies of ezetimibe + atorvastatin (10/80 mg) or ezetimibe + rosuvastatin (10/20 mg or 10/40 mg); non-statin lipid-lowering agents including fish oils containing >900 mg/day of eicosapentaenoic acid and docosahexaenoic acid (EPA+DHA), red yeast extract, Cholestin™, bile acid sequestrants, other cholesterol-lowering agents, niacin (>200 mg/day), or fibrates; systemic corticosteroids; psyllium, other fiber-based laxatives, phytosterol margarines, and/or over the counter (OTC) therapies known to affect serum lipid levels; orlistat or other anti-obesity medications and not maintained on a stable dose; any cyclical hormones; warfarin treatment without a stable dose or a stable International Normalized Ratio (INR).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

REFERENCES:
- [Result] Bays HE, Chen E, Tomassini JE, McPeters G, Polis AB, Triscari J. Fixed-dose combination ezetimibe+atorvastatin lowers LDL-C equivalent to co-administered components in randomized trials: use of a dose-response model. Fundam Clin Pharmacol. 2015 Apr;29(2):209-18. doi: 10.1111/fcp.12096. Epub 2015 Feb 27. PMID 25431239

RESULTS

PARTICIPANT FLOW:
Groups:
- Co-administration/Combination Sequence: Co-administration Ezetimibe 10 mg and Atorvastatin 40 mg then Ezetimibe/Atorvastatin 10 mg/40 mg fixed-dose combination
- Combination/Co-administration Sequence: Ezetimibe/Atorvastatin 10 mg/40 mg fixed-dose combination then Co-administration Ezetimibe 10 mg and Atorvastatin 40 mg
Period: Period 1
Arm/Group | Co-administration/Combination Sequence | Combination/Co-administration Sequence
Started | 164 | 164
Completed | 150 | 154
Not Completed | 14 | 10
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 5 | 5
Period: Crossover Washout
Arm/Group | Co-administration/Combination Sequence | Combination/Co-administration Sequence
Started | 150 | 154
Completed | 141 | 150
Not Completed | 9 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Non-compliance with Study Drug | 0 | 2
Period: Period 2
Arm/Group | Co-administration/Combination Sequence | Combination/Co-administration Sequence
Started | 141 | 150
Completed | 138 | 146
Not Completed | 3 | 4
Not completed — Adverse Event | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-administration/Combination Sequence | Combination/Co-administration Sequence | Total
Number analyzed (Participants) | 164 | 164 | 328
Age, Customized [Number; unit: Participants]
  30 to 39 years | 10 | 9 | 19
  40 to 49 years | 35 | 29 | 64
  50 to 59 years | 74 | 61 | 135
  60 to 64 years | 20 | 35 | 55
  ≥ 65 years | 25 | 30 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 92 | 186
  Male | 70 | 72 | 142

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) After 6 Weeks of Treatment
Description: Serum LDL-C calculated using Friedewald formula at baseline and after 6 weeks of treatment in each of the 2 treatment periods.
Time Frame: Baseline and Week 6
Population: Per-Protocol (PP) population, which excluded participants due to important deviations from the protocol that may have substantially affected the results of the primary efficacy endpoint(s). A participant may have been a protocol violator in 1 treatment period and not in the other treatment period.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Groups:
- Ezetimibe/Atorvastatin Fixed Dose Combination: Ezetimibe/atorvastatin 10 mg/40 mg combination tablet once daily for 6 weeks
- Co-Administration Ezetimibe and Atorvastatin: Ezetimibe 10 mg co-administered with atorvastatin 40 mg once daily for 6 weeks
Arm/Group | Ezetimibe/Atorvastatin Fixed Dose Combination | Co-Administration Ezetimibe and Atorvastatin
Number analyzed (Participants) | 280 | 280
Percentage Change | -58.9 [-60.9 to -56.9] | -58.7 [-60.7 to -56.7]
Statistical Analysis 1: Comparison: Ezetimibe/Atorvastatin Fixed Dose Combination vs Co-Administration Ezetimibe and Atorvastatin; It was anticipated that 85% of the enrolled participants would be evaluable to achieve 95% power in order to establish equivalence between the Ezetimibe/Atorvastatin Fixed Dose Combination and the co-administration of Ezetimibe and Atorvastatin with respect to percent change from baseline in LDL-C after 6 weeks of treatment using two one-sided tests each at 2.5% α-level, assuming the underlying true treatment difference is ±1.08% and that the standard deviation of the difference is 12.8%; Test type: Non-Inferiority or Equivalence — Equivalence was declared if the 97.5% expanded confidence interval for the mean difference between the fixed-dose combination and co-administration in percent change from baseline was contained within ±4%; ANCOVA; Difference in Least-squares means = -0.2, 97.5% CI 2-sided [-1.9 to 1.4]

2. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) After 6 Weeks of Treatment
Description: Serum TC measured at baseline and after 6 week of treatment in each of the 2 treatment periods.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe/Atorvastatin Fixed Dose Combination | Co-Administration Ezetimibe and Atorvastatin
Number analyzed (Participants) | 280 | 280
Percentage Change | -43.0 [-44.5 to -41.5] | -42.9 [-44.4 to -41.4]
Statistical Analysis 1: Comparison: Ezetimibe/Atorvastatin Fixed Dose Combination vs Co-Administration Ezetimibe and Atorvastatin; Test type: Superiority or Other; ANCOVA; Difference in Least-squares means = -0.1, 97.5% CI 2-sided [-1.4 to 1.2]

3. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) After 6 Weeks of Treatment
Description: Serum HDL-C measured at baseline and after 6 weeks of treatment in each of the 2 treatment periods.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe/Atorvastatin Fixed Dose Combination | Co-Administration Ezetimibe and Atorvastatin
Number analyzed (Participants) | 280 | 280
Percentage Change | 2.3 [0.8 to 3.8] | 2.6 [1.2 to 4.1]
Statistical Analysis 1: Comparison: Ezetimibe/Atorvastatin Fixed Dose Combination vs Co-Administration Ezetimibe and Atorvastatin; Test type: Superiority or Other; ANCOVA; Difference in Least-squares means = -0.3, 97.5% CI 2-sided [-1.8 to 1.2]

4. Secondary Outcome: Percent Change From Baseline in Non-high-density Lipoprotein Cholesterol (Non-HDL-C) After 6 Weeks of Treatment
Description: Non-HDL-C calculated at baseline and after 6 weeks of treatment in each of the 2 treatment periods.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe/Atorvastatin Fixed Dose Combination | Co-Administration Ezetimibe and Atorvastatin
Number analyzed (Participants) | 280 | 280
Percentage Change | -55.4 [-57.2 to -53.5] | -55.2 [-57.0 to -53.4]
Statistical Analysis 1: Comparison: Ezetimibe/Atorvastatin Fixed Dose Combination vs Co-Administration Ezetimibe and Atorvastatin; Test type: Superiority or Other; ANCOVA; Difference in Least-squares Means = -0.2, 97.5% CI 2-sided [-1.7 to 1.4]

5. Secondary Outcome: Percent Change From Baseline in Apolipoprotein (Apo) B After 6 Weeks of Treatment
Description: Serum Apo B measured at baseline and after 6 weeks of treatment in each of the 2 treatment periods.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe/Atorvastatin Fixed Dose Combination | Co-Administration Ezetimibe and Atorvastatin
Number analyzed (Participants) | 278 | 279
Percentage Change | -48.7 [-50.4 to -47.0] | -48.3 [-50.0 to -46.6]
Statistical Analysis 1: Comparison: Ezetimibe/Atorvastatin Fixed Dose Combination vs Co-Administration Ezetimibe and Atorvastatin; Test type: Superiority or Other; ANCOVA; Difference in Least-squares means = -0.5, 97.5% CI 2-sided [-1.9 to 1.0]

6. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) After 6 Weeks of Treatment
Description: Serum TG measured at baseline and after 6 weeks of treatment in each of the 2 treatment periods.
Time Frame: Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Ezetimibe/Atorvastatin Fixed Dose Combination | Co-Administration Ezetimibe and Atorvastatin
Number analyzed (Participants) | 280 | 280
Percentage Change | -36.2 [-40.4 to -31.6] | -36.2 [-38.8 to -33.5]
Statistical Analysis 1: Comparison: Ezetimibe/Atorvastatin Fixed Dose Combination vs Co-Administration Ezetimibe and Atorvastatin; Test type: Superiority or Other; constrained Longitudinal Data Analysis; Difference in Least-squares Means = 0.0, 97.5% CI 2-sided [-4.9 to 4.9]

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: All Patients as Treated Population defined as all randomized participants who received at least 1 dose of study drug. Adverse events were reported by actual treatment regardless of study period or assigned treatment sequence. Not all
  randomized participants entered Period 2 and therefore did not receive their assigned crossover treatment.
Groups:
- Co-Administration Ezetimibe and Atorvastatin: Ezetimibe 10 mg co-administered with atorvastatin 20 mg once daily for 6 weeks
Arm/Group | Ezetimibe/Atorvastatin Fixed Dose Combination | Co-Administration Ezetimibe and Atorvastatin
Serious Adverse Events (participants affected / at risk) | 3/303 | 2/313
Other Adverse Events (participants affected / at risk) | 0/303 | 0/313
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe/Atorvastatin Fixed Dose Combination (N=303) | Co-Administration Ezetimibe and Atorvastatin (N=313)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.